CLINICAL TRIAL: NCT04840771
Title: Optical Cohrence Tomography Angiography as a New Predictive Biomarker in Anatomical and Functional Recovery After Endoscopic Endonasal Pituitary Surgery: a Prospective Study
Brief Title: Predictive OCTA Biomarkers After Endoscopic Endonasal Pituitary Surgery
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 04/21
Record Dates: First submitted 2021-04-04; First posted 2021-04-12 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Endonasal Pituitary Surgery — Surgical treatment consisted of an endoscopic endonasal approach using a rigid 0-degree endoscope, 18 cm in length and 4 mm in diameter.

SUMMARY:
This study evaluates the structural parameters, by spectral domain optical coherence tomography (OCT), retinal vessel density, using OCT angiography, and visual acuity in patients that received endoscopic endonasal approach for the removal of an intra-suprasellar pituitary adenoma compressing the optic nerve.

DETAILED DESCRIPTION:
The primary outcome was to detect the changes in visual acuity, retinal structural and vascular features at 48 hours and 1 year after Endoscopic Endonasal Approach for the removal of an intra-suprasellar pituitary adenoma compressing the optic nerve.

The secondary outcome was to identify potential biomarker that could predict the functional recovery at 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* age older than 40 years
* diagnosis of pituitary adenoma
* treatment-naïve with Endoscopic Endonasal Pituitary Surgery
* absence of other neurological diseases
* absence of vitreoretinal and vascular retinal diseases

Exclusion Criteria:

* age younger than 40 years
* No diagnosis of pituitary adenoma
* previous treatments with Endoscopic Endonasal Pituitary Surgery
* presence of neurological diseases
* presence of vitreoretinal and vascular retinal diseases

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participans were older than 4 years with pituitary adenoma. They did not present other ophthalmological and neurological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Comparison between retinal structures before and 48 hours and 1 year after Endoscopic Endonasal Pituitary Surgery | 48 hours and 1 year follow up
  8 patients with pituitary adenoma compressing optic chiasm. Changes in thickness of ganglion cell complex (microns) and in thickness of retinal nerve fiber layer (microns) before and 48 hours and 1 year after Endoscopic Endonasal Pituitary Surgery
Comparison between retinal microvasculature before and 48 hours and 1 year after Endoscopic Endonasal Pituitary Surgery | 48 hours and 1 year follow up
  8 patients with pituitary adenoma compressing optic chiasm. Changes in retinal vessel density (percent) in macular and papillary regions before and 48 hours and 1 year after Endoscopic Endonasal Pituitary Surgery

SECONDARY OUTCOMES:
Correlation between retinal structures and visual acuity after Endoscopic Endonasal Pituitary Surgery | 1 year follow up
  8 patients with pituitary adenoma compressing optic chiasm underwent Endoscopic Endonasal Pituitary Surgery.
  Correlation between ganglion cell complex, retinal nerve fiber layer thicknesses (microns) at baseline and visual acuity recovery (logMAR) 1 year after surgery.
Correlation between retinal microvasculature and visual acuity after Endoscopic Endonasal Pituitary Surgery | 1 year follow up
  8 patients with pituitary adenoma compressing optic chiasm underwent Endoscopic Endonasal Pituitary Surgery.
  Correlation between retinal vessel density (percent) at baseline and visual acuity recovery (logMAR) 1 year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy